CLINICAL TRIAL: NCT07186608
Title: Specific Dietary Fibers May Enhance Colonic Adaptation in Short Bowel Syndrome (SBS) Through Microbial and Metabolic Mechanisms That Drive Functional Compensation.
Brief Title: Specific Dietary Fibers May Enhance Colonic Adaptation in Short Bowel Syndrome Through Microbial and Metabolic Mechanisms That Drive Functional Compensation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Wang Xinying, Chief Physician, Jinling Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20250918
Record Dates: First submitted 2025-09-19; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Select the party or parties who are masked (blinded) in the clinical study. If there is no masking, (Experimental)
  Interventions: Dietary Supplement: Dietary fiber intervention

INTERVENTIONS:
Dietary Supplement: Dietary fiber intervention — Ten patients with short bowel syndrome in clinical practice were subjected to dietary fiber intervention. Blood and fecal samples were collected before and after the dietary fiber intervention, and nutritional and intestinal barrier-related indicators were also collected to observe the improvement effect of dietary fiber on these patients.

SUMMARY:
Ten patients with short intestines in clinical practice were intervened with dietary fiber. Serum and feces before and after the dietary fiber intervention were collected, and relevant indicators of nutrition and intestinal barrier were collected to observe the improvement of dietary fiber on patients with short intestines

ELIGIBILITY:
All participants in Cohort 1 were recruited at the Eastern Theatre Command General Hospital (Nanjing, China) and provided written informed consent. The primary inclusion criterion was a confirmed diagnosis of type II or type III short bowel syndrome in patients aged 18

-70 years. Participants were excluded if they had other gastrointestinal diseases, malignant tumours, autoimmune diseases, infectious diseases or renal insufficiency (severe kidney disease with creatinine levels exceeding 3.0 mg/dL), or if they had taken antibiotics for more than three days within the preceding three months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Determination of nitrogen content | From enrollment to the end of treatment at 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Theater Command General Hospital, Nanjing, China